CLINICAL TRIAL: NCT01306279
Title: The Infective Pulmonary Exacerbations in Cystic Fibrosis - an Ecological Perspective
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 11/H0713/7
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Infection; Pulmonary exacerbation; Hypermutators; Bacterial diversity; Quorum sensing
MeSH Terms: conditions — Cystic Fibrosis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cystic Fibrosis, infection: Cystic Fibrosis patients with an infective exacerbation

SUMMARY:
Given the treatment burden and excess morbidity and mortality associated with acute infective exacerbations in cystic fibrosis, a clear understanding of the mechanisms involved in the origins of an infective exacerbation and the response to antibiotics is vital to improving long-term outcomes in CF.

This study will examine 3 areas of interest in CF exacerbations.

1. Bacterial biodiversity and its clinical significance
2. The role of bacteria which are able to rapidly mutate (hypermutators)
3. Inter-bacterial communication and its role in infective exacerbations

Study Hypothesis 1

Increased microbiological diversity represents a balanced community of bacteria. The presence of a diverse population of bacteria in CF infections therefore predicts a better outcome for treatment than when a population consists of a small number of more virulent organisms.

Study Hypothesis 2

Pseudomonas aeruginosa hypermutators can mutate much more often than ordinary Pseudomonas aeruginosa bacteria. Hypermutators are likely to grow better when the bacteria are under stress, such as during antibiotic treatment or during an infection. They are, however, weaker organisms because of the multiple mutations they have undergone. Their presence does not relate to clinical outcome but may be associated with the emergence of antibiotic resistance.

Study Hypothesis 3

Some Pseudomonas aeruginosa bacteria communicate with each other by secreting and responding to chemicals known as quorum sensing (QS)molecules. As well as affecting the behaviour of bacteria, these QS molecules can cause inflammation in the lung of CF patients. Selective growth of QS-producing organisms can trigger lung exacerbations in CF. If antibiotics kill this population of bacteria and QS molecule levels drop in the lung, patients recover from infection quickly. Failure to kill these bacteria with antibiotics allow QS molecule levels to remain elevated and patients to have prolonged infections.

DETAILED DESCRIPTION:
We will sequentially recruit patients attending our CF centre with an infective exacerbation of CF, who are chronically infected with Pseudomonas aeruginosa.

We will record spirometry, blood markers of inflammation, quality of life questionnaires and investigate sputum samples for:

1. Routine microbiology
2. Bacterial diversity using 16s RNA identification techniques
3. Relative abundance of P.aeruginosa hypermutators
4. Levels of quorum sensing molecules

These observations will be undertaken before commencing intravenous antibiotic therapy, on days 7, 10 and the last day of antibiotic therapy. Patients will also be reviewed one month after the end of antibiotic therapy where spirometry and a sputum sample will be collected for the above investigations.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Cystic Fibrosis
* Chronic Pseudomonas aeruginosa
* Symptoms and signs of infective exacerbation

Exclusion Criteria:

* age under 16
* unable to give consent or patients with significant mental health problems
* co-existent active allergic bronchopulmonary aspergillosis requiring a change in steroid or antifungal therapy
* a previous participant in this study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with Cystic Fibrosis attending to commence intravenous antibiotics for a pulmonary exacerbation of CF
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Hodson, MD MSc FRCP, Principal Investigator — Imperial College London
Locations (1):
- Department of Cystic Fibrosis, NHLI, Imperial College,, London, London, United Kingdom